CLINICAL TRIAL: NCT00375713
Title: A Multi-centre, Double-blind, Double-dummy, Randomized, Active-controlled Phase III Study to Evaluate the Efficacy and Safety of Xyzal® 5mg od vs Zyrtec® 10mg od in Subjects Aged 15 Years and Above With Dermatitis and Eczema
Brief Title: Randomized Phase III Study to Evaluate the Efficacy and Safety of Xyzal® (Levocetirizine) vs Zyrtec® (Cetirizine) in Subjects With Dermatitis and Eczema
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: UCB Pharma (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: A00410
Record Dates: First submitted 2006-09-12; First posted 2006-09-13 (Estimated); Results first posted 2009-10-14 (Estimated); Last update posted 2011-08-31 (Estimated); Status verified 2009-12

CONDITIONS: Dermatitis; Eczema
Keywords: Dermatitis; Eczema; Pruritus; Xyzal; Zyrtec; Levocetirizine; Cetirizine
MeSH Terms: conditions — Dermatitis; Eczema; Pruritus | interventions — levocetirizine; Cetirizine; Hydrocortisone; Ointments

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Levocetirizine (Experimental): Levocetirizine + Cetirizine-Placebo + Standard Topical Steroid (1% hydrocortisone) Ointment for 14 days
  Interventions: Drug: Levocetirizine; Drug: Placebo-Cetirizine; Drug: Standard topical steroid (1% hydrocortisone) ointment
- Cetirizine (Active Comparator): Cetirizine + Levocetirizine-Placebo + Standard Topical Steroid (1% hydrocortisone) Ointment for 14 days
  Interventions: Drug: Cetirizine; Drug: Placebo-Levocetirizine; Drug: Standard topical steroid (1% hydrocortisone) ointment

INTERVENTIONS:
Drug: Levocetirizine — 1 Levocetirizine 5mg tablet per day before bedtime for 14 days
  Other Names: Xyzal®
  Arms: Levocetirizine
Drug: Cetirizine — 1 Cetirizine 10mg tablet per day before bedtime for 14 days.
  Other Names: Zyrtec®
  Arms: Cetirizine
Drug: Placebo-Levocetirizine — 1 Placebo-Levocetirizine tablet per day before bedtime for 14 days
  Arms: Cetirizine
Drug: Placebo-Cetirizine — 1 Placebo-Cetirizine tablet per day before bedtime for 14 days
  Arms: Levocetirizine
Drug: Standard topical steroid (1% hydrocortisone) ointment — 1% hydrocortisone ointment, applied 2-3 times a day to all affected areas

SUMMARY:
Korean double-blind non-inferiority study to asses the efficacy (as measured by the responder rate of pruritus severity score by the patient at visit 4 or end-of-treatment visit over the 2 weeks treatment period) and safety of Xyzal® to Zyrtec® in subjects suffering from dermatitis and eczema with pruritus symptoms

ELIGIBILITY:
Inclusion Criteria:

* Subjects diagnosed as having atopic dermatitis, contact dermatitis, prurigo, pruritus in the dermatitis and eczema
* Subjects who require and agree to the concomitant use of a topical steroid preparation.
* Subjects having a minimum level of pruritus and having used topical hydrocortisone during the run -in period
* Written informed consent signed and dated by subject/legal guardian
* Female subjects with childbearing potential are eligible if they use a medically accepted contraceptive method and have a negative pregnancy test.

Exclusion Criteria:

* Subjects with a known hypersensitivity to cetirizine or levocetirizine
* Any clinically significant condition that might interfere with the treatment evaluation, both for efficacy and safety
* Have used forbidden concomitant medications or having not respected adequate wash-out periods as defined by the protocol

Min Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 466 (Actual)
Dates: Start 2005-10; Primary Completion 2006-05 (Actual); Study Completion 2006-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kevin Beh, MD, Study Director — UCB Pharma
Locations (3):
- South Korea (3):
  - Gyeunggi-do
  - Kyeonggi-Do
  - Seoul

REFERENCES:
- See also: FDA Safety Alerts and Recalls — http://www.fda.gov/Safety/MedWatch/SafetyInformation/default.htm

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 506 patients were screened and 466 randomized. Due to a packaging error 99 patients were excluded from the efficacy analysis according to the advice of the Korean FDA. The Reported Adverse Events section refers to the Safety Population (N= 423) defined as all patients treated with at least one safety evaluation without entry criteria violation.
Pre-assignment Details: Participant workflow refers to all randomized subjects whereas in Baseline Characteristics numbers and statistics for the modified Intent To Treat (m-ITT) population are presented (see definition of m-ITT population in the Outcome Measure section).
Groups:
- Levocetirizine: Levocetirizine 5 mg tablet once daily plus Placebo - Cetirizine 10 mg tablet once daily plus standard topical steroid ointment
- Cetirizine: Cetirizine 10 mg tablet once daily plus Placebo - Levocetirizine 5 mg once daily plus standard topical steroid ointment
Period: Overall Study
Arm/Group | Levocetirizine | Cetirizine
Started | 232 (Randomized population (N=232).) | 234 (Randomized population (N=234).)
Completed | 212 (20 Patients were not treated or discontinued after randomization in Levocetirizine group.) | 211 (23 Patients were not treated or discontinued after randomization in Cetirizine group.)
Not Completed | 20 | 23

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Levocetirizine | Cetirizine | Total
Number analyzed (Participants) | 168 | 172 | 340
Age Continuous [Mean (Standard Deviation); unit: years] | 30.17 (10.09) | 30.11 (10.60) | 30.14 (10.34)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 113 | 120 | 233.0
  Male | 55 | 52 | 107.0
Region of Enrollment [Number; unit: participants]
  Korea, Republic of | 168 | 172 | 340

OUTCOME MEASURES:

1. Primary Outcome: Responder Status According to Pruritus Severity Score (Response = Mild or None in Pruritus Severity Score).
Description: A participant is a responder if the pruritus severity score is assessed as mild or none, otherwise it is a non-responder. The responder status is defined at day 14, except if the investigator assessed the subject as a responder at day 7. The Pruritus Score is in general defined as: 3 for Severe, 2 for Moderate, 1 for Mild and 0 for None.
Time Frame: Day 7 and 14
Population: The modified ITT population is defined as all randomized patients who received the study drug, except the patients who did not meet the entry criteria, took prohibited medication during the study period, did not have any available data for efficacy evaluation and who were enrolled with packing errors.
Measure: Number; unit: Participants
Arm/Group | Levocetirizine | Cetirizine
Number analyzed (Participants) | 168 | 172
Participants
  Responder | 131 | 134
  Non-Responder | 37 | 38
Statistical Analysis 1: Comparison: Levocetirizine vs Cetirizine; The lower bound of the 95% two sided confidence interval for the difference (Levocetirizine - Cetirizine) in percentage of responders is compared to the pre-set threshold for non inferiority (-10% which is equal to -0.1 for the proportion of responders). Standard method for estimation of the difference in proportions incl. confidence interval using normal approximation is used; Test type: Non-Inferiority or Equivalence — The pre-set threshold for non inferiority is -10%; Difference in proportion of responders = 0.00069213, 95% CI [-0.0875 to 0.0888]

2. Secondary Outcome: Change From Baseline in the Mean Pruritus Severity Score at Endpoint During the 14 Day Treatment Period
Description: The Pruritus Score Scale ranges from 0 to 3 (3 for Severe, 2 for Moderate, 1 for Mild and 0 for None). Endpoint is at visit 4 on day 14 or at an earlier timepoint at study completion.
Time Frame: Baseline and at endpoint during the 14 day treatment period
Population: All patients in modified Intent-to-treat population. Last Observation Carried Forward principle was applied to the missing data of the pruritus severity score on the previous day of the randomization.
Measure: Mean (Standard Error); unit: Units on a scale
Arm/Group | Levocetirizine | Cetirizine
Number analyzed (Participants) | 168 | 172
Units on a scale | 1.15 (0.05) | 1.21 (0.05)
Statistical Analysis 1: Comparison: Levocetirizine vs Cetirizine; The mean daily pruritus score at Day 14 visit or at study completion was analyzed using an analysis of covariance (ANCOVA) model, including pruritus severity score of the day before the randomization as a covariate and treatment group as a factor; Test type: Superiority or Other; p = 0.4369, ANCOVA; Pruritus score is adjusted on pruritus Baseline score

3. Secondary Outcome: Duration of Pruritus (Stated in Categories) at Endpoint During the 14 Day Treatment Period
Description: Duration of pruritus was categorized as follows: 3 if > 6 hours/24hr, 2 if 1 to 6 hours/24hr, 1 if less than 1 hour/24hr, and 0 if No pruritus. The endpoint is visit 4 on day 14 or at an earlier time point at study completion.
Time Frame: At endpoint during the 14 day treatment period
Population: as for outcome 2
Measure: Mean (Standard Error); unit: Units on a scale
Arm/Group | Levocetirizine | Cetirizine
Number analyzed (Participants) | 168 | 172
Units on a scale | 2.13 (0.05) | 2.20 (0.05)
Statistical Analysis 1: Comparison: Levocetirizine vs Cetirizine; The categorized duration of Pruritus at endpoint during the 14 day treatment period was analyzed using an analysis of covariance (ANCOVA) model, including pruritus severity score of the day before the randomization as a covariate and treatment group as a factor; Test type: Superiority or Other; p = 0.3549, ANCOVA; pruritus severity score at baseline has been used as a covariate

4. Secondary Outcome: Global Improvement at Endpoint During the 14 Day Treatment Period
Description: Global improvement is measured on an ordered nominal scale ranging from marked improvement to exacerbation (see categories in the table). The endpoint is visit 4 on day 14 or at an earlier time point at study completion.
Time Frame: At endpoint during the 14 day treatment period
Population: All patients in modified ITT except 1 patient in levocetirizine group and 3 patients in cetirizine group who have missing values.
Measure: Number; unit: Participants
Arm/Group | Levocetirizine | Cetirizine
Number analyzed (Participants) | 167 | 169
Participants
  Marked improvement | 47 | 52
  Moderate improvement | 62 | 54
  Mild improvement | 39 | 47
  No change | 18 | 15
  Exacerbation | 1 | 1
Statistical Analysis 1: Comparison: Levocetirizine vs Cetirizine; Test type: Superiority or Other; p = 0.7518, Cochran-Mantel-Haenszel; stratified on the prurity severity score at the previous day of randomization

ADVERSE EVENTS:
Arm/Group | Levocetirizine | Cetirizine
Serious Adverse Events (participants affected / at risk) | 1/209 | 0/214
Other Adverse Events (participants affected / at risk) | 0/209 | 5/214
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Levocetirizine (N=209) | Cetirizine (N=214)
Leukemia acute (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Levocetirizine (N=209) | Cetirizine (N=214)
Rhinitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 5 (5)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
UCB has > 60 days but <= 180 days to review results communications prior to public release and may delete information that compromises ongoing studies or is considered proprietary. This restriction is not intended to compromise the objective scientific integrity of the manuscript, it being understood that results shall be published regardless of outcome.